CLINICAL TRIAL: NCT07347691
Title: Predicting Atrial Fibrillation in Patients With Post-implantable Cardiac Monitor Implementation : A Prospective, Long-term Follow-up Study Using Comprehensive AI ECG Analysis : Multicenter Prospective Study
Brief Title: AI-Based Prediction of Atrial Fibrillation in ESUS Patients With ICM
Acronym: SMART-ESUS
Status: Recruiting | Type: Observational
Sponsor: Inha University Hospital (Other)
Collaborators: DeepCardio Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yong-Soo Baek, Professor, Inha University Hospital
Other Study IDs: 2024-07-024
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Implantable Cardiac Monitor; Artificial Intelligence; Deep Learning; Electrocardiography; Risk Prediction; Cryptogenic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk Group: Patients classified as having a high risk of atrial fibrillation by the SmartECG-AF AI algorithm.
- Low to Intermediate Risk Group: Patients classified as having a low to intermediate risk of atrial fibrillation by the SmartECG-AF AI algorithm.

SUMMARY:
This study investigates patients with Embolic Stroke of Undetermined Source (ESUS) who have received an Implantable Cardiac Monitor (ICM). The main purpose is to evaluate the predictive value of an Artificial Intelligence ECG analysis tool, named SmartECG-AF.

Participants will be classified into two groups based on the AI analysis: a "High Risk" group and a "Low to Intermediate Risk" (control) group. The study aims to compare the incidence rate of atrial fibrillation (AF) events over time between these two groups. Additionally, the study will analyze the relationship between the AI-predicted risk levels and the occurrence of major cardiovascular events during the follow-up period.

DETAILED DESCRIPTION:
Embolic Stroke of Undetermined Source (ESUS) accounts for a significant proportion of ischemic strokes, and occult Atrial Fibrillation (AF) is considered a major etiology. While Implantable Cardiac Monitors (ICMs) are the gold standard for long-term rhythm monitoring, identifying patients at the highest risk for AF remains a clinical challenge.

This multicenter, prospective study aims to validate the clinical utility of an artificial intelligence-based electrocardiogram analysis algorithm, "SmartECG-AF," in this specific population. The algorithm analyzes 12-lead ECGs recorded during sinus rhythm to detect subtle signs of electrical remodeling associated with paroxysmal AF.

Enrolled patients with ESUS who have undergone ICM implantation will have their baseline ECGs analyzed by the SmartECG-AF algorithm. Based on the AI-generated probability score, patients will be stratified into a "High Risk" group and a "Low to Intermediate Risk" group. The study will longitudinally track these patients to compare the time-to-event for ICM-detected AF between the two groups. Additionally, the study will evaluate the correlation between the AI risk score and the incidence of Major Adverse Cardiovascular Events (MACE), providing evidence for AI-guided risk stratification in cryptogenic stroke management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 years or older.
* Patients diagnosed with Embolic Stroke of Undetermined Source (ESUS) who have undergone or are scheduled for Implantable Cardiac Monitor (ICM) implantation.
* Patients who have undergone at least one 12-lead ECG examination within 2 weeks before or after the date of ICM implantation.
* Patients maintaining Sinus Rhythm on ECG at the time of enrollment.
* Patients who have voluntarily signed the informed consent form.

Exclusion Criteria:

* Patients diagnosed with Atrial Fibrillation (AF) at least once prior to the date of enrollment.
* Patients whose ICM battery status is at Elective Replacement Interval (ERI), making recording impossible.
* Patients whose ECGs cannot be analyzed by the AI algorithm (SmartECG-AF) due to severe artifacts or noise, or are incompatible with digital analysis.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Embolic Stroke of Undetermined Source (ESUS) aged 30 years or older who have received or are scheduled to receive an Implantable Cardiac Monitor (ICM). Participants are recruited from five tertiary referral hospitals in South Korea (Inha University Hospital, Jeju National University Hospital, Korea University Guro Hospital, Korea University Ansan Hospital, and Ajou University Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Atrial Fibrillation (Time-to-Event) | Up to 12 months
  Comparison of the cumulative incidence rate of atrial fibrillation (AF) events between the High Risk group and the Low to Intermediate Risk group (classified by SmartECG-AF). AF occurrence is confirmed by reviewing data recorded on the Implantable Cardiac Monitor (ICM).

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | Up to 12 months
  Evaluation of the composite rate of major clinical events including recurrent stroke, hospitalization for heart failure, myocardial infarction, and all-cause death (cardiovascular and non-cardiovascular). The study will analyze the correlation between the occurrence of these events and the AI-predicted risk levels.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Soo Baek, MD, PhD, Principal Investigator — Inha University Hospital
Locations (5):
- South Korea (5):
  - Korea University Ansan Hospital, Ansan
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality. The informed consent form signed by participants does not include authorization for the release of individual raw data to third parties.